CLINICAL TRIAL: NCT03836612
Title: Healthcare Resource Utilisation, Common Mental Health Problems, and Infections in People With Inflammatory Bowel Disease (IBD)
Brief Title: Healthcare Resource Utilisation, Common Mental Health Problems, and Infections in People With Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: Momentum Data (Industry)
Collaborators: Pfizer (Industry); University of Surrey (Other)
Responsible Party: Sponsor
Other Study IDs: P003
Record Dates: First submitted 2019-01-17; First posted 2019-02-11 (Actual); Results first posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2021-10

CONDITIONS: Inflammatory Bowel Diseases; Ulcerative Colitis; Crohn Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People with inflammatory bowel disease: Adults (18+) with inflammatory bowel disease registered with a contributing GP practice during the study period
  Interventions: Other: No intervention
- Controls: Adults (18+) without inflammatory bowel disease registered with a contributing GP practice during the study period
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observation of routine clinical practice

SUMMARY:
Ulcerative colitis and Crohn's disease are the commonest types of inflammatory bowel disease (IBD). Both conditions range in severity from no symptoms to being potentially fatal. Both conditions are treated with medications which suppress the immune system. It is not known whether this increases the risk for infections and cancers in these conditions. It is also recognised by healthcare professionals that these conditions cause a considerable amount of psychological distress. However, this has never been measured in a large population sample.

This study will investigate any associations with treatment and new onset infections and cancer. They will also examine the relationship between IBD and common mental health problems (specifically, depression and anxiety) and the impact that these have on the healthcare use (including number of general practitioner [GP] appointments, hospital attendances, and medication prescriptions. Combined, these studies should provide a better understanding of the impact of IBD on affected people and provide evidence to support the correct allocation of healthcare resources.

DETAILED DESCRIPTION:
Objective We aim to provide an accurate and contemporary measurement of the current healthcare resource utilisation in people with inflammatory bowel disease (IBD); namely ulcerative colitis (UC) and Crohn's disease (CD). We also aim to provide estimates of infection incidence in this population and the prevalence of common mental health conditions.

Method We will identify UC and CD using algorithms validated for accurately identifying these conditions from primary care records in the United Kingdom (UK). We will identify a prevalent cohort of adults with IBD with the Royal College of General Practitioners (RCGP) Research and Surveillance Centre (RSC) network over the last decade. We will identify a matched cohort of people without IBD; matched on age, gender and primary care practice. Across these cohorts we will compare healthcare resource utilisation (primary care attendances, number of primary care prescriptions for antidepressant and anxiolytic medications, number of primary care prescriptions for medications used in IBD, recorded secondary care attendances, and issue of statements of fitness for work), incident infections (any common infection, any viral infection, or any gastrointestinal infection), and common mental health conditions (depression and anxiety).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years over the study period
* Registered with a contributing primary care practice for any duration during the study period

Exclusion Criteria:

* IBD not classifiable or of a type other than UC or Crohn's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All individuals with an existing or incident diagnosis of UC or CD during the study period (2013-2018), defined by the presence of at least one disease-specific diagnostic code will be eligible for inclusion in the IBD cohort. Controls will matched people without IBD matched on age, gender and primary care practice.
Sampling Method: Non-Probability Sample
Enrollment: 95055 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew McGovern, MD, Study Director — Momentum Data Ltd
Locations (1):
- Momentum Data Ltd, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data (IPD) is confidential but can be made available in an anonymised form to bone fide researchers subject to the required data protection training and other requirements. All data will remain behind a firewall and will only be available for access through a secured computer network.
Supporting Information: Study Protocol
Time Frame: There is no pre-specified time-frame for data availability; this will be considered on an individual basis for each request.
Access Criteria: As above

REFERENCES:
- [Derived] Irving P, Barrett K, Tang D, Nijher M, de Lusignan S. Common infections, mental health problems and healthcare use in people with inflammatory bowel disease: a cohort study protocol. Evid Based Ment Health. 2021 May;24(2):82-87. doi: 10.1136/ebmental-2020-300167. Epub 2020 Sep 17. PMID 32943436

RESULTS

PARTICIPANT FLOW:
Groups:
- People With Inflammatory Bowel Disease (Cases): Adults (18+) with inflammatory bowel disease registered with a contributing General Practitioner (GP) practice during the study period
  No intervention: Observation of routine clinical practice
- People Without Inflammatory Bowel Disease (Controls): Adults (18+) without inflammatory bowel disease registered with a contributing GP practice during the study period
  No intervention: Observation of routine clinical practice
Period: Overall Study
Arm/Group | People With Inflammatory Bowel Disease (Cases) | People Without Inflammatory Bowel Disease (Controls)
Started | 19011 | 76044
Completed | 19011 | 76044
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- People With Inflammatory Bowel Disease (Cases): Adults (18+) with inflammatory bowel disease registered with a contributing GP practice during the study period
  No intervention: Observation of routine clinical practice
- Total: Total of all reporting groups
Arm/Group | People With Inflammatory Bowel Disease (Cases) | People Without Inflammatory Bowel Disease (Controls) | Total
Number analyzed (Participants) | 19011 | 76044 | 95055
Age, Customized [Count of Participants; unit: Participants]
  18-29 | 2276 | 9416 | 11692
  30-39 | 3036 | 11931 | 14967
  40-49 | 3379 | 13593 | 16972
  50-59 | 3560 | 14305 | 17865
  60-69 | 3235 | 12890 | 16125
  70-79 | 2278 | 8942 | 11220
  80+ | 1247 | 4967 | 6214
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9968 | 39746 | 49714
  Male | 9043 | 36298 | 45341
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 19011 | 76044 | 95055
BMI [Count of Participants; unit: Participants]
  Underweight (≤18.5) | 7229 | 24690 | 31919
  Normal weight (18.5-25) | 639 | 1814 | 2453
  Overweight (25-30) | 5824 | 23707 | 29531
  Obese (≥30) | 3775 | 17379 | 21154
  Not recorded | 1544 | 8454 | 9998
Index of Multiple Deprivation (IMD) quintile [Count of Participants; unit: Participants]
  1 (most deprived) | 2396 | 9933 | 12329
  2 | 2846 | 11514 | 14360
  3 | 3617 | 14720 | 18337
  4 | 4684 | 18137 | 22821
  5 (least deprived) | 5117 | 20388 | 25505
  Not recorded | 351 | 1352 | 1703
Comorbidities - Type 2 diabetes [Count of Participants; unit: Participants] | 1665 | 6336 | 8001
Comorbidities - Hypertension [Count of Participants; unit: Participants] | 4249 | 17591 | 21840
Comorbidities - Atrial fibrillation [Count of Participants; unit: Participants] | 658 | 2336 | 2994
Comorbidities - Angina [Count of Participants; unit: Participants] | 606 | 2075 | 2681
Comorbidities - Myocardial infarction [Count of Participants; unit: Participants] | 481 | 1650 | 2131
Comorbidities - Stroke [Count of Participants; unit: Participants] | 387 | 1382 | 1769
Comorbidities - Heart failure [Count of Participants; unit: Participants] | 296 | 1062 | 1358
Comorbidities - Chronic liver disease [Count of Participants; unit: Participants] | 386 | 487 | 873
Comorbidities - Dementia [Count of Participants; unit: Participants] | 694 | 2786 | 3480
Comorbidities - Rheumatoid arthritis [Count of Participants; unit: Participants] | 281 | 706 | 987
Comorbidities - Asthma [Count of Participants; unit: Participants] | 3796 | 12924 | 16720
Comorbidities - Chronic Obstructive Pulmonary Disease (COPD) [Count of Participants; unit: Participants] | 982 | 2990 | 3972
Use of systemic therapy [Count of Participants; unit: Participants] | 4183 | 700 | 4883

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Anxiety Episodes (Crohn's Disease)
Description: Compare the prevalence of anxiety episodes in people with and without Crohn's disease.
  Number of people with at least one anxiety episode in people.
Time Frame: Measured over five years - 2014 to 2018 inclusive
Population: Subset of people diagnosed with IBD having Crohn's disease
Measure: Count of Participants; unit: Participants
Groups:
- People With Crohn's Disease (Cases): People aged ≥18, registered with a GP practice contributing to the Oxford-Royal College of General Practitioners Research and Surveillance Centre database (RCGP RSC) between 1 January 2014 and 1 January 2019 with an existing or incident diagnosis of Crohn's disease.
- People Without Crohn's Disease (Controls): People aged ≥18, registered with a GP practice contributing to the RCGP RSC between 1 January 2014 and 1 January 2019 without a history of IBD and matched with an individual with IBD.
Arm/Group | People With Crohn's Disease (Cases) | People Without Crohn's Disease (Controls)
Number analyzed (Participants) | 7557 | 30228
Participants | 262 | 892

2. Primary Outcome: Prevalence of Anxiety Episodes (Ulcerative Colitis)
Description: Compare the prevalence of anxiety episodes in people with and without Ulcerative Colitis.
  Number of people with at least one anxiety episode
Time Frame: Measured over five years - 2014 to 2018 inclusive
Population: Subset of people diagnosed with IBD having Ulcerative Colitis
Measure: Count of Participants; unit: Participants
Groups:
- People With Ulcerative Colitis (Cases): People aged ≥18, registered with a GP practice contributing to the RCGP RSC between 1 January 2014 and 1 January 2019 with an existing or incident diagnosis of Ulcerative Colitis.
- People Without Ulcerative Colitis (Controls): People aged ≥18, registered with a GP practice contributing to the RCGP RSC between 1 January 2014 and 1 January 2019 without a history of IBD and matched with an individual with IBD.
Arm/Group | People With Ulcerative Colitis (Cases) | People Without Ulcerative Colitis (Controls)
Number analyzed (Participants) | 11454 | 45816
Participants | 341 | 1221

3. Primary Outcome: Prevalence of Depressive Episodes (Crohn's Disease)
Description: Compare the prevalence of depressive episodes in people with and without Crohn's disease.
  Number of people with at least one depressive episode
Time Frame: Measured over five years - 2014 to 2018 inclusive
Population: Subset of people diagnosed with IBD having Crohn's disease
Measure: Count of Participants; unit: Participants
Groups:
- People With Crohn's Disease (Cases): People aged ≥18, registered with a GP practice contributing to the RCGP RSC between 1 January 2014 and 1 January 2019 with an existing or incident diagnosis of Crohn's disease.
Arm/Group | People With Crohn's Disease (Cases) | People Without Crohn's Disease (Controls)
Number analyzed (Participants) | 7557 | 30228
Participants | 431 | 1233

4. Primary Outcome: Prevalence of Depressive Episodes (Ulcerative Colitis)
Description: Compare the prevalence of depressive episodes in people with and without Ulcerative Colitis.
  Number of people with at least one depressive episode.
Time Frame: Measured over five years - 2014 to 2018 inclusive
Population: Subset of people diagnosed with IBD having Ulcerative Colitis
Measure: Count of Participants; unit: Participants
Arm/Group | People With Ulcerative Colitis (Cases) | People Without Ulcerative Colitis (Controls)
Number analyzed (Participants) | 11454 | 45816
Participants | 507 | 1666

5. Primary Outcome: Number of People With Depressive Disorder in People With and Without Crohn's Disease
Description: Compare the prevalence of depressive disorder in people with and without Crohn's disease.
Time Frame: Measured over five years - 2014 to 2018 inclusive
Population: Subset of people diagnosed with IBD having Crohn's disease
Measure: Count of Participants; unit: Participants
Arm/Group | People With Crohn's Disease (Cases) | People Without Crohn's Disease (Controls)
Number analyzed (Participants) | 7557 | 30228
Participants | 1322 | 3911

6. Primary Outcome: Number of People With Depressive Disorder in People With and Without Ulcerative Colitis
Description: Compare the prevalence of depressive disorder in people with and without Ulcerative Colitis.
Time Frame: Measured over five years - 2014 to 2018 inclusive
Population: Subset of people diagnosed with IBD having Ulcerative colitis
Measure: Count of Participants; unit: Participants
Arm/Group | People With Ulcerative Colitis (Cases) | People Without Ulcerative Colitis (Controls)
Number analyzed (Participants) | 11454 | 45816
Participants | 1627 | 5676

7. Primary Outcome: Number of People With at Least One Infection Event in Those With and Without Ulcerative Colitis
Description: Number of people with at least one infection event during follow up for any common infection, gastrointestinal infection, and any viral infection.
Time Frame: Measured over 5 years - 2014 to 2018 inclusive
Measure: Count of Participants; unit: Participants
Groups:
- People With Ulcerative Colitis (Common Infections Cases): People aged ≥18, registered with a GP practice contributing to the RCGP RSC between 1 January 2014 and 1 January 2019 with an existing or incident diagnosis of Ulcerative Colitis.
- People Without Ulcerative Colitis (Common Infections Controls): People aged ≥18, registered with a GP practice contributing to the RCGP RSC between 1 January 2014 and 1 January 2019 without a history of Ulcerative Colitis and matched with an individual with Ulcerative Colitis.
Arm/Group | People With Ulcerative Colitis (Common Infections Cases) | People Without Ulcerative Colitis (Common Infections Controls)
Number analyzed (Participants) | 11360 | 45440
Participants
  Any common infection | 5111 | 17403
  Gastrointestinal infection | 510 | 1365
  Viral infection | 2544 | 8510

8. Primary Outcome: Number of People With at Least One Infection Event in Those With and Without Crohn's Disease
Description: as for outcome 7
Time Frame: Measured over 5 years - 2014 to 2019 inclusive
Measure: Count of Participants; unit: Participants
Groups:
- People With Crohn's Disease (Common Infections Cases): People aged ≥18, registered with a GP practice contributing to the RCGP RSC between 1 January 2014 and 1 January 2019 with an existing or incident diagnosis of Crohn's disease.
- People Without Crohn's Disease (Common Infections Controls): People aged ≥18, registered with a GP practice contributing to the RCGP RSC between 1 January 2014 and 1 January 2019 without a history of Crohn's disease and matched with an individual with Crohn's disease.
Arm/Group | People With Crohn's Disease (Common Infections Cases) | People Without Crohn's Disease (Common Infections Controls)
Number analyzed (Participants) | 7469 | 29876
Participants
  Any common infection | 3470 | 11227
  Gastrointestinal infection | 395 | 841
  Viral infection | 1797 | 5917

9. Primary Outcome: Number of People With at Least One Sub-infection Event in Those With and Without Ulcerative Colitis
Description: Sub-infection outcomes: Upper respiratory tract infection (URTI), Pneumonia, Acute Bronchitis, Influenza, Skin infection, Genital infection, urinary tract infection (UTI), GI infection subset (only stool culture confirmed Clostridium difficile, Salmonella, Shigella, and Campylobacter infections), Herpes Simplex infection, Herpes Zoster infection
Time Frame: Measured over 5 years - 2014 to 2019 inclusive
Measure: Count of Participants; unit: Participants
Arm/Group | People With Ulcerative Colitis (Common Infections Cases) | People Without Ulcerative Colitis (Common Infections Controls)
Number analyzed (Participants) | 11360 | 45440
Participants
  URTI | 2118 | 7143
  Pneumonia | 100 | 288
  Acute Bronchitis | 1754 | 5554
  Influenza | 234 | 856
  Skin infections | 1654 | 5268
  Genital infection | 246 | 874
  UTI | 733 | 2631
  GI infection subset | 121 | 198
  Herpes Simplex infection | 106 | 352
  Herpes Zoster infection | 309 | 839

10. Secondary Outcome: Healthcare Resource Utilization - Primary Care Visits
Description: Compare healthcare resource utilization in people with and without IBD, and stratifying by IBD type and compare healthcare resource utilization in people with IBD, with and without mental health illness.
Time Frame: Measured over five years - 2014 to 2018 inclusive
Population: The arm/Groups titled people with ulcerative colitis and people with Crohn's disease are subsets of the arm/Group titled people with IBD
Measure: Number (95% Confidence Interval); unit: Visits per person per year
Groups:
- People With IBD: People aged ≥18, registered with a GP practice contributing to the RCGP RSC between 1 January 2014 and 1 January 2019 with an existing or incident diagnosis of Crohn's disease or ulcerative colitis.
- People With Ulcerative Colitis: People aged ≥18, registered with a GP practice contributing to the RCGP RSC between 1 January 2014 and 1 January 2019 with an existing or incident diagnosis of ulcerative colitis.
- People With Crohn's Disease: People aged ≥18, registered with a GP practice contributing to the RCGP RSC between 1 January 2014 and 1 January 2019 with an existing or incident diagnosis of Crohn's disease.
- People Without IBD: People aged ≥18, registered with a GP practice contributing to the RCGP RSC between 1 January 2014 and 1 January 2019 without a history of IBD.
Arm/Group | People With IBD | People With Ulcerative Colitis | People With Crohn's Disease | People Without IBD
Number analyzed (Participants) | 19011 | 11454 | 7557 | 76044
Visits per person per year | 6.41 [6.39 to 6.44] | 6.18 [6.15 to 6.20] | 6.78 [6.75 to 6.82] | 4.49 [4.48 to 4.50]

11. Secondary Outcome: Healthcare Resource Utilization - Secondary Care Emergency Attendances
Description: as for outcome 10
Time Frame: Measured over five years - 2014 to 2018 inclusive
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Attendances per person per year
Arm/Group | People With IBD | People With Ulcerative Colitis | People With Crohn's Disease | People Without IBD
Number analyzed (Participants) | 19011 | 11454 | 7557 | 76044
Attendances per person per year | 0.455 [0.449 to 0.461] | 0.396 [0.389 to 0.403] | 0.546 [0.536 to 0.557] | 0.259 [0.257 to 0.262]

12. Secondary Outcome: Healthcare Resource Utilization - Fitness for Work Notes
Description: as for outcome 10
Time Frame: Measured over five years - 2014 to 2018 inclusive
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Notes issued per person per year
Arm/Group | People With IBD | People With Ulcerative Colitis | People With Crohn's Disease | People Without IBD
Number analyzed (Participants) | 19011 | 11454 | 7557 | 76044
Notes issued per person per year | 0.311 [0.306 to 0.316] | 0.270 [0.265 to 0.276] | 0.378 [0.368 to 0.386] | 0.215 [0.213 to 0.217]

13. Secondary Outcome: Healthcare Resource Utilization: Medications for Mental Health Conditions - Selective Serotonin Reuptake Inhibitors (SSRIs)
Description: as for outcome 10
Time Frame: Measured over five years - 2014 to 2018 inclusive
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Prescriptions per person per year
Arm/Group | People With IBD | People With Ulcerative Colitis | People With Crohn's Disease | People Without IBD
Number analyzed (Participants) | 19011 | 11454 | 7557 | 76044
Prescriptions per person per year | 1.328 [1.317 to 1.338] | 1.218 [1.205 to 1.230] | 1.495 [1.478 to 1.512] | 1.046 [1.041 to 1.050]

14. Secondary Outcome: Healthcare Resource Utilization: Medications for Mental Health Conditions - Anxiolytic Medications
Description: as for outcome 10
Time Frame: Measured over five years - 2014 to 2018 inclusive
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Prescriptions per person per year
Arm/Group | People With IBD | People With Ulcerative Colitis | People With Crohn's Disease | People Without IBD
Number analyzed (Participants) | 19011 | 11454 | 7557 | 76044
Prescriptions per person per year | 0.219 [0.214 to 0.223] | 0.189 [0.183 to 0.194] | 0.264 [0.257 to 0.272] | 0.166 [0.164 to 0.168]

15. Primary Outcome: Number of People With at Least One Sub-infection Event in Those With and Without Crohn's Disease
Description: Sub-infection outcomes: URTI, Pneumonia, Acute Bronchitis, Influenza, Skin infection, Genital infection, UTI, GI infection subset (only stool culture confirmed Clostridium difficile, Salmonella, Shigella, and Campylobacter infections), Herpes Simplex infection, Herpes Zoster infection
Time Frame: Measured over 5 years - 2014 to 2019 inclusive
Measure: Count of Participants; unit: Participants
Arm/Group | People With Crohn's Disease (Common Infections Cases) | People Without Crohn's Disease (Common Infections Controls)
Number analyzed (Participants) | 7469 | 29876
Participants
  URTI | 1475 | 5002
  Pneumonia | 59 | 136
  Acute Bronchitis | 1059 | 3211
  Influenza | 158 | 621
  Skin infections | 1201 | 3294
  Genital infection | 219 | 665
  UTI | 473 | 1568
  GI infection subset | 76 | 130
  Herpes Simplex infection | 109 | 253
  Herpes Zoster infection | 237 | 491

ADVERSE EVENTS:
Description: Death, serious adverse events and other (non-serious adverse events) were not assessed for the study.
Arm/Group | People With Inflammatory Bowel Disease (Cases) | People Without Inflammatory Bowel Disease (Controls)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/12/NCT03836612/Prot_SAP_000.pdf